CLINICAL TRIAL: NCT05304390
Title: Tailoring Screening and Smoking Cessation for the LGBTQ Community
Brief Title: A Tailored Screening and Smoking Cessation Program for the LGBTQ Community of Seattle
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to end of funding. Enrollment sufficient to evaluate primary and secondary outcomes measures.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: LUNGevity Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1122073; NCI-2022-01427 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10815 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-03-08; First posted 2022-03-31 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Patient Navigation; Smoking Devices; Carbon Monoxide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health services research (patient navigation intervention) (Experimental): Participants receive a patient navigation intervention consisting of a series of points of contact (mostly via telephone) between the PN/TTS and includes: 1) An introduction and enrollment in LCS, 2) facilitation of a SDM visit with the LCS-dedicated nurse practitioner, 3) individual assessment of barriers and facilitators to in-person low-dose CT screening, 4) explanation of results and needed follow-up, and 5) follow-up reminders. Participants also undergo carbon monoxide measurement by exhaling into a disposable monitor for 10 seconds at the initial visit and the post-intervention visit. The PN may also provide an intervention for smoking cessation.
  Interventions: Behavioral: Patient Navigation; Other: Questionnaire Administration; Behavioral: Smoking Cessation Intervention; Procedure: Carbon Monoxide Measurement

INTERVENTIONS:
Behavioral: Patient Navigation — Receive patient navigation intervention
  Other Names: Patient Navigator Program
Other: Questionnaire Administration — Ancillary studies
Behavioral: Smoking Cessation Intervention — Receive an intervention for smoking cessation
  Other Names: Smoking and Tobacco Use Cessation Interventions
Procedure: Carbon Monoxide Measurement — Undergo carbon monoxide measurement
  Other Names: CMONOX

SUMMARY:
This clinical trial develops a tailored screening and smoking cessation program for the lesbian, gay, bisexual, transgender (trans) and queer (LGBTQ) community of Seattle, Washington. A lung cancer screening program may help LGTBQ people who smoke overcome unique barriers that keep them from receiving preventive care, and constantly facing healthcare discrimination. Members of the LGBTQ community have historically smoked at higher rates than the general population and thus could benefit greatly from targeted efforts to improve lung cancer screening and smoking cessation implementation.

DETAILED DESCRIPTION:
OUTLINE:

AIM 1: Stakeholders (community organization leaders, medical providers of LGBTQ patients, and LGBTQ community members and tobacco users) participate in an interview over 45 minutes to 1 hour.

AIM 2: Participants participate in focus groups over 1-1.5 hours.

AIM 3: Participants receive a patient navigation intervention consisting of a series of points of contact (mostly via telephone) between the patient navigator/tobacco treatment specialist (PN/TTS) and includes: 1) An introduction and enrollment in LCS, 2) facilitation of a shared decision-making (SDM) visit with the LCS-dedicated nurse practitioner, 3) individual assessment of barriers and facilitators to in-person low-dose CT screening, 4) explanation of results and needed follow-up, and 5) follow-up reminders. Participants also undergo carbon monoxide measurement by exhaling into a disposable monitor for 10 seconds at the initial visit and the post-intervention visit. The PN may also provide an intervention for smoking cessation.

After completion of Aim 3 study intervention, participants are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1 MEDICAL PROVIDER OF LGBTQ PATIENTS: Age minimum of 18
* AIM 1 MEDICAL PROVIDER OF LGBTQ PATIENTS: Affiliation with Cancer Consortium, Seattle's LGBTQ Center, or other organization serving LGBTQ persons
* AIM 1 MEDICAL PROVIDER OF LGBTQ PATIENTS: Identifies as providing primary care or specialty care to largely LGBTQ population (doctor of medicine [MD], registered nurse [RN], physician assistants [PA], advanced registered nurse practitioner [ARNP])
* AIM 1, COMMUNITY ORGANIZATION LEADERS: Age minimum of 18
* AIM 1, COMMUNITY ORGANIZATION LEADERS: Broadly defined as "community leader" (i.e. leadership in Seattle-area volunteer, philanthropic, community service groups) in discussions with with community-based participatory research (CBPR) partners
* AIM 2: Current cigarette smoker (defined as actively smoking within the last 6 months, this is consistent with (c/w) standard and Seattle Cancer Care Alliance (SCCA) definition of "current smoker") or former cigarette smoker
* AIM 2: Aged 50-80 years
* AIM 2: At least 20 pack-year smoking history
* AIM 3: Identify as a member of the LGBTQ community
* AIM 3: Eligible for no-cost sharing LCS based on United States Preventive Services Task Force (USPSTF) criteria

  * As of Jan 2022: aged 50-80 years, at least 20 pack-year smoking history, and currently smoke tobacco cigarettes [as this intervention is based around current cigarette smokers (as defined above)], former cigarette smokers not included in this Aim

Exclusion Criteria:

* AIM 1: Non-English speaking participants
* AIM 2: Those found to be ineligible for LCS on coordinator review; or who are non-English speaking or have cognitive dysfunction that would prevent participation in SDM
* AIM 3: Those found to be ineligible for LCS on coordinator review; or who are non-English speaking or have cognitive dysfunction that would prevent participation in SDM

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Number of lesbian, gay, bisexual, transgender (trans) and queer (LGBTQ) community stakeholders who participate in the Aim 1 interviews/focus groups (Aim 1) | Up to 3 months
Number of LBGTQ community members who participate in the Aim 2 focus groups (Aim 2) | Up to 9 months
Acceptability of patient navigation and smoking cessation interventions (Aim 3) | Up to 12 months
  The Acceptability of Intervention Measure (AIM) will be summarized and presented as range of scores from 1 (low acceptability) to 5 (high acceptability), with at least 75% of participants giving the interventions at least a "4", the threshold for acceptability.
Patient satisfaction with navigator throughout navigation and smoking cessation interventions (Aim 3) | Up to 12 months
  The Patient Satisfaction with Navigator (PSN-1) will also be summarized and presented as range of scores from 1 (high satisfaction) to 5 (low satisfaction), with at least 75% of participants giving the navigator interactions at maximum a "2", the threshold for satisfaction.
Effectiveness of navigation visit(s): knowledge (Aim 3) | Up to 12 months
  Pre- and post-intervention Lung cancer screening Knowledge Survey (LKS) responses will be compared via Cochran-Mantel-Haenszel tests for all categorical data.
Effectiveness of navigation visit(s): smoking cessation (Aim 3) | Up to 12 months
  Initiation of pharmacotherapy and/or behavioral treatment, floating cigarette abstinence (>7 days abstinence among those currently smoking at intervention start date, as defined in post-intervention survey) [Aim 3]

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Triplette, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Triplette M, Omernik B, Snidarich M, Heffner JL, Brooks E, Crothers K, Brown MC, Murphy NR, Louie T. Tailored Patient Navigation to Support Lung Cancer Screening and Smoking Cessation in LGBTQ+ Individuals: A Pilot Study. Ann Am Thorac Soc. 2025 Oct;22(10):1592-1600. doi: 10.1513/AnnalsATS.202502-215OC. PMID 40440319

DOCUMENTS (1):
  • Informed Consent Form (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT05304390/ICF_000.pdf